CLINICAL TRIAL: NCT00789789
Title: Cohort Study of Volunteers That Have Participated to Preventive HIV-1 Vaccine Trials
Status: Terminated | Type: Observational
Why Stopped: stopped prematurely due to the absence of safety signal
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2007-002219-14; ANRS COV1 COHVAC
Record Dates: First submitted 2008-11-10; First posted 2008-11-13 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: HIV Infection; HIV Seronegativity
Keywords: Cohort; HIV uninfected volunteers; HIV preventive vaccine; Long term safety
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimen collection (serum, plasma and whole blood)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1

SUMMARY:
This cohort study should provide an exhaustive overview on long-term safety of various preventive HIV-vaccines administered in phase I and II clinical trials to healthy volunteers of the ANRS network.

DETAILED DESCRIPTION:
Since 1992, 16 phase I and II clinical trials have been performed by the French National Agency for Research on AIDS and Viral Hepatitis (ANRS) evaluating the safety of several HIV-1 vaccine candidates and their capacity to induce immune responses. The ANRS program has evaluated a recombinant HIV-1 envelope protein Rgp-160, canarypox ALVAC vectors, and mixtures of lipopeptides whose sequences represent CTL-epitopes of HIV-1 Gag, Pol and Nef proteins. Most of them have been administered intramuscularly but recently, mucosal immunization and intradermal route were used. Previously compiled in a published meta-analysis, safety studies were restricted to the duration of the trials.

ANRS establishes a cohort study in order to describe the long-term safety of preventive HIV-vaccines administered in phase I and II clinical trials to healthy volunteers of the "ANRS volunteer-network" in France and to gather clinical and biological data in a database and blood specimen collection which could be analysed in case of a long-term safety issue in ANRS vaccine trials or if pertinent, in other HIV vaccine trials ANRS COV1-COHVAC is a prospective, multicentric cohort study composed of participants in preventive HIV-vaccines phase I and II trials. All ANRS volunteers who ever received one dose of a candidate vaccine are eligible and those who are going to complete their participation to a clinical trial during the cohort study time.

The ANRS COV1-COHVAC project relies on a long-term follow-up of the cohort (at least 7 years after the end of the vaccine trial), that includes the retrospective and prospective collection of medical and biological data [severe health events (grade 3-4), as well as neurological, ophtalmological, and immunological events (any grade), starting from the first injection of a candidate vaccine, are recorded], blood specimen collections and psycho-behavioral evaluations (self-questionnaires and interviews) in order to collect data about consequences of participation and experience of possible HIV vaccine-induced seropositivity in such trials.

Of the ANRS "volunteer-network", 206 participants have been involved in the early trials and are actually eligible to participate in this cohort. Altogether with the more recent studies completed or in progress, the cohort will comprise at least 400 individuals in 2009.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers of the "ANRS volunteer network" who have received at least one dose of a vaccine candidate in a HIV preventive clinical trial.
* volunteers who have signed an informed consent

Exclusion Criteria:

* volunteers not covered by Health Insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 488 (Actual)
Dates: Start 2008-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Description of severe health events (grade 3-4), as well as neurological, ophtalmological, and immunological events (any grade), starting from the first injection of a HIV candidate vaccine. | once a year

SECONDARY OUTCOMES:
Evaluation of HIV serologic status by two ELISA tests and Western blot test ( only if ELISA is positive). | once a year
Evaluation of psycho-behavioral consequences, associated to participation in a HIV preventive trial, on entourage, familial, professional and social relations, with a self-questionnaire and an interview with a clinician. | once a year
Incidence of HIV infection (frequency, description of contamination). | once a year

CONTACTS AND LOCATIONS:
Overall Officials: Odile LAUNAY, MD, PhD, Principal Investigator — CIC Cochin Pasteur, Hôpital Cochin, Paris, France; Laurence MEYER, MD, PhD, Study Chair — INSERM SC-10-US019, Villejuif, France
Locations (1):
- CIC Cochin Pasteur, hôpital Cochin, Paris, France